CLINICAL TRIAL: NCT03487341
Title: Placental Cord Drainage After Vaginal Delivery: A Randomized Clinical Trial
Brief Title: Placental Cord Drainage After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AS1751
Record Dates: First submitted 2018-03-24; First posted 2018-04-04 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cord drainage (Active Comparator)
  Interventions: Other: Cord drainage
- Cord clamping (Active Comparator)
  Interventions: Other: Cord clamping

INTERVENTIONS:
Other: Cord drainage — Cord drainage
  Arms: Cord drainage
Other: Cord clamping — Cord clamping
  Arms: Cord clamping

SUMMARY:
Placental Cord Drainage after Vaginal Delivery A randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Pregnancy with vertex presentation.
* Gestational age37 up to 42 weeks
* Patient expected to have spontaneous vaginal delivery.
* Maternal age 18 years old or more.

Exclusion Criteria:

* Previous history of Postpartum hemorrhage.
* Antepartum hemorrhage
* Multiple pregnancies
* Instrumental deliveries
* Coagulation disorders
* Over distended uterus (hydramnios, large fetus).
* Patient with extensive extended vaginal or cervical tear.
* Rupture uterus.
* Secondary arrest of cervical dilatation.
* Persistent occipito-posterior.
* Deep transverse arrest of fetal head.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
blood loss | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt